CLINICAL TRIAL: NCT01075646
Title: Randomised and Double-blind Clinical Trial on Post-operative Analgesic Efficacy in Colorectal Surgery and Hepatic Surgery With Continuous Infusion of Local Anesthesia vs Saline Serum in the Surgical Incision.
Brief Title: Local Anesthesia Versus Saline Serum in Surgical Incision of Colorectal or Hepatic Surgery
Acronym: CATROP-2007
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, antonia dalmau llitjos, MD PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANESTHESIA SERVICE HUB
Record Dates: First submitted 2010-01-11; First posted 2010-02-25 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Postoperative Pain; Surgery; Postoperative Complications
Keywords: postoperative pain; wound infusion; local anesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Experimental): After a bolus administration of Ropivacaine a perfusion ot the same anesthetic is initiated through an elastomeric wound during 48 hours
  Interventions: Drug: ropivacaine
- saline solution (Placebo Comparator): After a bolus administration of saline solution a perfusion ot saline solution is initiated through an elastomeric wound during 48 hours
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: ropivacaine — Laparotomy of colorectal surgery: 10 ml bolus ropivacaine 0,75% + infusion with elastomeric pump with ropivacaine 0,38% at a 5ml/h.
  Laparoscopy of colorectal surgery: 5 ml bolus ropivacaine 0,75% + infusion with elastomeric pump with ropivacaine 0,38% at a 2 ml/h.
  Hepatic surgery: 10 ml de ropivacaine 0,45% + infusion with elastomeric pump with ropivacaine 0,23 at a 5ml/h.
  Other Names: (wound infusion ropivacaine)
  Arms: Ropivacaine
Drug: saline solution — Laparotomy of colorectal surgery: 10 ml bolus saline solution 0.9% + infusion with elastomeric pump with saline solution 0.9% at a 5ml/h.
  Laparoscopy of colorectal surgery: 10 ml bolus saline solution 0.9% + infusion with elastomeric pump with saline solution 0.9% at a 2 ml/h.
  Hepatic surgery: 10 ml de saline solution 0.9% + infusion with elastomeric pump with saline solution 0.9% at a 5ml/h
  Other Names: wound infusion saline solution
  Arms: saline solution

SUMMARY:
The purpose of this study is to determine whether a continuous infusion of local anesthesia with a catheter in the surgical wound reduces patient consumption of opiates by 30% in the 48-hour postoperative period following surgery for colorectal neoplasm and hepatic surgery versus the continuous infusion of physiological serum.

DETAILED DESCRIPTION:
Postoperative analgesia in major abdominal surgery is managed with intravenous PCA (patient controlled analgesia) with morphine associated to non-steroidal anti-inflammatories drugs (NSAD) and paracetamol in the first 48 hours of the postoperative phase. With this multimodal approach patients undergoing colorectal surgery have a median pain score on the verbal scale (0-10) of 3 (range 0-8) with a mean of morphine consumption of 54 mg (SD 24 mg) and patients undergoing hepatic surgery have a median pain score of 2(range 0-7) with a mean of morphine consumption of 28 mg (SD 17 mg).

Although opiates are very potent analgesics they also produce side effects and numerous studies have demonstrated a significant reduction in morbidity when patients received lower dose of opiates during anesthesia and in postoperative period. Continuous infusion of local anesthetics in the surgical wound has been used for pain control in different types of surgeries. However, controversial reports has been reported in abdominal surgery.

We are conducting prospective, randomised and double-blind placebo control trials in two surgical models (colo-rectal oncologic surgery and hepatic resection) using continuous perfusion of ropivacaine 0.38% in the surgical wound versus saline.

Anesthetic protocol is the same for all patients.

Patients undergoing colo-rectal surgery can be operated either in laparotomy or laparoscopic technique therefore patients are stratified into four groups once surgical closure has begun:

* Group A1 ropivacaine and laparotomy
* Group A2 ropivacaine and laparoscopy
* Group B1 saline and laparotomy
* Group B2 saline and laparoscopy

In the preanesthesia visit patients who match inclusion criteria are invited to participate in the study and they signed the informed consent. When the patient is in the theatre a nurse not involved in the management of patients opens a closed envelope which indicates the solution to be prepared according to the assigned group.

The surgeon inserts a multiperforated catheter at the subfascial level of surgical wound , just below the suture of the muscular fascia (between the peritoneum and the muscular fascia) and after that surgeons finish the subcutaneous plane and the skin. After the closure a bolus of 5 ml (laparoscopy colon surgery)or 10 ml (laparotomy colon and hepatic surgery) of the solution is given through the catheter and subsequently an elastomer filled with ropivacaine or saline is connected. The catheter is fixed to the skin with steri-strip and sterile dressing.

During the procedure we administer in a protocol basis the NSAD and thirty minutes before the end of the surgery we administer morphine. In the postoperative period the patient receives a NSAD regime and a PCA morphine treatment.

The catheter is withdrawn after 48 hours and also the PCA and the analgesic treatment is with NSAD.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Undergoing scheduled colorectal cancer and hepatic surgery
* Patients must be able to understand the PCA (the self administration system)

Exclusion Criteria:

* Background of allergic reaction or contraindication for local anesthesia or non steroid anti-inflammatory drugs.
* Patient with epidural catheter or receiving combined analgesia during surgery (age above 80, moderate-severe respiratory dysfunction, patients who prior presented complex postoperative pain management.
* Emergency surgery
* Patients with risk of hepatic insufficiency (Klatskin's tumor, extended right hepatectomy, right hepatectomy in patients with steatosis, hepatic resection in patients over 70 years of age who have been given chemotherapy).
* Inflammatory bowel disease: ulcerative colitis, Crohn's disease.
* Major psychiatric condition.
* Patients with active drug addiction or on chronic treatment with opiates.
* Morbid obesity (BMI > 35 kg/m2)
* Patients with heart disease (myocardiopathy, conduction alterations, antiarrhythmic treatment) and severe liver disease (alteration synthesis, histolysis and or cholestasis).
* Patients with kidney failure.
* Patients treated with fluvoxamine (antidepressant) and enoxacin (antibiotic) both are potent inhibitors of CYPIA2.
* Septic patients
* Patients that do not wish to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2009-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antònia Dalmau Llitjós, Physical D, Study Director — Univeritary Hospital of Bellvitge. IDIBELL
Locations (1):
- Anesthesiology Service of Univeritary Hospital of Bellvitge, Hospitalet . Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu SS, Richman JM, Thirlby RC, Wu CL. Efficacy of continuous wound catheters delivering local anesthetic for postoperative analgesia: a quantitative and qualitative systematic review of randomized controlled trials. J Am Coll Surg. 2006 Dec;203(6):914-32. doi: 10.1016/j.jamcollsurg.2006.08.007. Epub 2006 Oct 25. No abstract available. PMID 17116561
- [Background] Beaussier M, El'Ayoubi H, Schiffer E, Rollin M, Parc Y, Mazoit JX, Azizi L, Gervaz P, Rohr S, Biermann C, Lienhart A, Eledjam JJ. Continuous preperitoneal infusion of ropivacaine provides effective analgesia and accelerates recovery after colorectal surgery: a randomized, double-blind, placebo-controlled study. Anesthesiology. 2007 Sep;107(3):461-8. doi: 10.1097/01.anes.0000278903.91986.19. PMID 17721249
- [Background] Wu CL, Partin AW, Rowlingson AJ, Kalish MA, Walsh PC, Fleisher LA. Efficacy of continuous local anesthetic infusion for postoperative pain after radical retropubic prostatectomy. Urology. 2005 Aug;66(2):366-70. doi: 10.1016/j.urology.2005.02.030. PMID 16040091
- [Background] Gupta A, Perniola A, Axelsson K, Thorn SE, Crafoord K, Rawal N. Postoperative pain after abdominal hysterectomy: a double-blind comparison between placebo and local anesthetic infused intraperitoneally. Anesth Analg. 2004 Oct;99(4):1173-1179. doi: 10.1213/01.ANE.0000130260.24433.A2. PMID 15385371
- [Background] Zohar E, Fredman B, Phillipov A, Jedeikin R, Shapiro A. The analgesic efficacy of patient-controlled bupivacaine wound instillation after total abdominal hysterectomy with bilateral salpingo-oophorectomy. Anesth Analg. 2001 Aug;93(2):482-7, 4th contents page. doi: 10.1097/00000539-200108000-00048. PMID 11473884
- [Background] Fredman B, Zohar E, Tarabykin A, Shapiro A, Mayo A, Klein E, Jedeikin R. Bupivacaine wound instillation via an electronic patient-controlled analgesia device and a double-catheter system does not decrease postoperative pain or opioid requirements after major abdominal surgery. Anesth Analg. 2001 Jan;92(1):189-93. doi: 10.1097/00000539-200101000-00036. PMID 11133625
- [Background] Chester JF, Ravindranath K, White BD, Shanahan D, Taylor RS, Lloyd-Williams K. Wound perfusion with bupivacaine: objective evidence for efficacy in postoperative pain relief. Ann R Coll Surg Engl. 1989 Nov;71(6):394-6. PMID 2604350
- [Background] Baig MK, Zmora O, Derdemezi J, Weiss EG, Nogueras JJ, Wexner SD. Use of the ON-Q pain management system is associated with decreased postoperative analgesic requirement: double blind randomized placebo pilot study. J Am Coll Surg. 2006 Feb;202(2):297-305. doi: 10.1016/j.jamcollsurg.2005.10.022. PMID 16427556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment took place at the hospital Universitari de Bellvitge in Barcelona, Spain, from April 2010 to April 2012 in the case of colorrectal surgery. In hepatic surgery the study recruitment took place at the same hospital, from April 2010 to June 2014.
Pre-assignment Details: In colorrectal surgery 117 patients were assessed for elegibility. Of these 50 patients were excluded before randomization including 23 with exclusion criteria and 18 with a surgical or organization reason. In hepatic surgery 108 patients were assesed for eligibility, 9 patients were excluded with a surgical reason.
Groups:
- Ropivacaine Colorectal Surgery: After a bolus administration of Ropivacaine a perfusion ot the same anesthetic is initiated through an elastomeric wound during 48 hours
  ropivacaine: Laparotomy of colorectal surgery: 10 ml bolus ropivacaine 0,75% + infusion with elastomeric pump with ropivacaine 0,38% at a 5ml/h.
  Laparoscopy of colorectal surgery: 5 ml bolus ropivacaine 0,75% + infusion with elastomeric pump with ropivacaine 0,38% at a 2 ml/h.
- Saline Solution Colorectal Surgery: After a bolus administration of saline solution a perfusion ot saline solution is initiated through an elastomeric wound during 48 hours
  placebo: Laparotomy of colorectal surgery: 10 ml bolus saline solution 0.9% + infusion with elastomeric pump with saline solution 0.9% at a 5ml/h.
  Laparoscopy of colorectal surgery: 10 ml bolus saline solution 0.9% + infusion with elastomeric pump with saline solution 0.9% at a 2 ml/h.
- Ropivacaine Hepatic Surgery: After a bolus administration of Ropivacaine a perfusion ot the same anesthetic is initiated through an elastomeric wound during 48 hours Hepatic surgery: 10 ml of ropivacaine 0,45% + infusion with elastomeric pump with ropivacaine 0,23 at a 5ml/h.
- Saline Solution Hepatic Surgery: After a bolus administration of saline solution a perfusion ot saline solution is initiated through an elastomeric wound during 48 hours Hepatic surgery: 10 ml de saline solution 0.9% + infusion with elastomeric pump with saline solution 0.9% at a 5ml/h
Period: Overall Study
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Started | 33 | 34 | 53 | 46
Completed | 29 | 31 | 52 | 44
Not Completed | 4 | 3 | 1 | 2
Not completed — Lost to Follow-up | 4 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery | Total
Number analyzed (Participants) | 33 | 34 | 53 | 46 | 166
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [41 to 80] | 64.5 [18 to 78] | 63.62 [61.38 to 65.85] | 59.73 [56.54 to 62.92] | 62.96 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 14 | 17 | 52
  Male | 20 | 26 | 39 | 29 | 114
Hypertension [Number; unit: participants]
  Yes | 15 | 17 | 23 | 15 | 70
  No | 18 | 17 | 30 | 31 | 96
Diabetes [Number; unit: participants]
  Yes | 10 | 7 | 10 | 11 | 38
  No | 23 | 27 | 43 | 35 | 128
Antiplatelet drugs [Number; unit: participants]
  Yes | 5 | 4 | 3 | 1 | 13
  No | 28 | 30 | 50 | 45 | 153
Anemia [Number; unit: participants]
  Yes | 3 | 2 | 2 | 2 | 9
  No | 30 | 32 | 51 | 44 | 157
Stroke [Number; unit: participants]
  Yes | 3 | 1 | 2 | 2 | 8
  No | 30 | 33 | 51 | 44 | 158
Myocardial disease [Number; unit: participants]
  Yes | 1 | 0 | 2 | 2 | 5
  No | 32 | 34 | 51 | 44 | 161
Chronic respiratory insuficiency [Number; unit: participants]
  Yes | 6 | 0 | 1 | 0 | 7
  No | 27 | 34 | 52 | 46 | 159
Surgical procedure [Number; unit: participants]
  Right hemicolectomy | 7 | 5 | 0 | 0 | 12
  Left hemicolectomy | 14 | 15 | 0 | 0 | 29
  Total colectomy | 1 | 4 | 0 | 0 | 5
  Rectal resections | 11 | 10 | 0 | 0 | 21
  mayor hepatectomy | 0 | 0 | 22 | 17 | 39
  minor hepatectomy | 0 | 0 | 30 | 29 | 59
  radiofrequency | 0 | 0 | 1 | 0 | 1
Duration of surgery [Median (Inter-Quartile Range); unit: minutes] | 205 [80 to 410] | 225 [90 to 420] | 274.26 [254.95 to 293.58] | 263.57 [240.42 to 286.73] | 241.95 [80 to 420]
Size of incision [Median (Inter-Quartile Range); unit: cm] | 16.5 [4 to 40] | 17.5 [5 to 37] | 31.5 [29.19 to 33.82] | 29.67 [27.69 to 31.65] | 23.79 [4 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Mg of Morphine Consumption During 48 Hours Administered by Patient Controlled Analgesia System
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Number analyzed (Participants) | 29 | 31 | 52 | 44
mg | 23 [11.25 to 42.75] | 52 [24.5 to 64] | 24.63 [19.97 to 29.29] | 26.78 [21.7 to 31.85]

2. Secondary Outcome: Intensity of Pain Measured by Verbal Pain Scale.
Description: Verbal pain scale is a numeric measure of intensity pain, values range from 0 (no pain) to 10 (excruciating pain), Each patient rate the paín that feel with a number from 0 to 10.
Time Frame: At interval periods during 48 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Number analyzed (Participants) | 33 | 34 | 53 | 46
units on a scale
  Verbal numeric scale 0h after surgery | 1 [0 to 3] | 2.5 [0 to 6.5] | 2.75 [1.94 to 3.57] | 2.5 [1.63 to 3.37]
  Verbal numeric scale 6h after surgery | 2 [1 to 3] | 3 [1 to 4] | 1.72 [1.33 to 2.1] | 2.38 [1.81 to 2.95]
  Verbal numeric scale 12h after surgery | 2 [1 to 3] | 2 [1 to 2.75] | 1.45 [1.09 to 1.81] | 1.8 [1.22 to 2.38]
  Verbal numeric scale 24h after surgery | 2 [2 to 3] | 2 [1 to 3] | 1.64 [1.32 to 1.96] | 2 [1.44 to 2.56]
  Verbal numeric scale 48h after surgery | 2 [1 to 3] | 2 [1 to 2] | 1.62 [1.29 to 1.94] | 2.14 [1.59 to 2.68]

3. Secondary Outcome: Time Spent Sitting in a Chair, Deambulation, Solid Ingestion.
Time Frame: 7 Days (from Day 8-15)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Number analyzed (Participants) | 33 | 34 | 53 | 46
hours
  Sitting in the chair | 46 [24 to 48] | 48 [42 to 48] | 51.75 [45.5 to 58] | 43.2 [38.25 to 48.14]
  Deambulation | 72 [48 to 104] | 72 [69 to 96] | 81.2 [73.71 to 88.69] | 87.37 [70.97 to 103.77]
  Solid food intake | 96 [72 to 120] | 120 [72 to 158] | 88 [79.8 to 96.19] | 79.79 [64.25 to 95.34]

4. Secondary Outcome: Secondary Effects Due to Morphine: Nausea and Vomiting
Time Frame: during 48 hours
Measure: Number; unit: participants
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Number analyzed (Participants) | 33 | 34 | 53 | 46
participants
  Yes | 5 | 6 | 2 | 6
  No | 28 | 28 | 51 | 40

5. Secondary Outcome: Local Reaction in the Wound and Insertion Point of the Catheter (Inflammation Signs and Infection)
Time Frame: During 8-15 days
Measure: Number; unit: participants
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Number analyzed (Participants) | 33 | 34 | 53 | 46
participants
  Yes | 6 | 10 | 2 | 2
  No | 27 | 24 | 51 | 44

6. Secondary Outcome: Contamination of the Catheter (Microbiologist Analysis)
Time Frame: at 48 hours
Measure: Number; unit: participants
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Number analyzed (Participants) | 33 | 34 | 53 | 46
participants
  Yes | 6 | 4 | 2 | 2
  No | 27 | 30 | 51 | 44

ADVERSE EVENTS:
Time Frame: We collected all adverse events appeared in the hospitalary period
Arm/Group | Ropivacaine Colorectal Surgery | Saline Solution Colorectal Surgery | Ropivacaine Hepatic Surgery | Saline Solution Hepatic Surgery
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/53 | 0/46
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/53 | 0/46

LIMITATIONS AND CAVEATS:
A limitation of the study is the high number of recruited patients who were excluded before ranodmization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes